CLINICAL TRIAL: NCT02488525
Title: Prevention of Hemorrhage After Implantation of Mechanical Circulatory Support
Acronym: PHAM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: deficient inclusion
Sponsor: University Hospital, Lille (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015_06; 2015-001231-20 (EudraCT Number); PHRC-14-0469 (Other: Ministry of health, France)
Record Dates: First submitted 2015-07-01; First posted 2015-07-02 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
Keywords: Acquired Von Willebrand; Gastro-intestinal bleeding; LVAD
MeSH Terms: conditions — Heart Failure; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wilfactin (Experimental): Prophylactic treatment with Wilfactin after implantation of continuous-flow left ventricular assist device reduces the frequency of bleeding in comparison to the usual care.
  Interventions: Drug: Prophylactic treatment with Wilfactin
- Control (No Intervention): The control group will receive all treatments according to standard of care which does not include prophylactic administration of Wilfactin®

INTERVENTIONS:
Drug: Prophylactic treatment with Wilfactin — Prophylactic treatment with Wilfactin after implantation of continuous-flow left ventricular assist device reduces the frequency of bleeding in comparison to the usual care.
  Other Names: Prophylactic treatment with VWF factor concentrate
  Arms: Wilfactin

SUMMARY:
Main objective of the study is to demonstrate that a prophylactic treatment with VWF factor concentrate after implantation of continuous-flow left ventricular assist device (CF-LVAD) reduces the frequency of clinically significant bleeding within 3 months after implantation in comparison to the usual care. Adult patients with functional defects of VWF measured after implantation of continuous LVAD are randomly assigned to prophylactic treatment.

DETAILED DESCRIPTION:
This time point was chosen because the bleeding events are maximal within the first 3 months after implantation.

* Adult patients > 18 years who need a CF-LVAD due to advanced heart failure.
* Functional To determine the potential indication of Wilfactin® in the field of CF-LVAD and avoid widespread use and to establish evidence-based recommendation To improve the knowledge of the role of VWF concentrate in bleeding and angiogenesis after CF-LVAD implantation and to provide some results about mechanism involved angiogenesis or hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years who need a CF-LVAD due to advanced heart failure.
* Functional defects of VWF measured between day 2 and day 4 after implantation (either PFA-ADP closure time >180 sec and or VWF:Act/VWF:Ag≤ 0.7)
* Informed consent of the patient or support person in case of disability at baseline (patient intubated and ventilated)

Exclusion Criteria:

* Treatment with Wilfactin® within the last seven days
* Previous adverse reaction to Wilfactin®
* Absence of functional defects of VWF measured between day 2 and day 4 after implantation (either PFA-ADP closure time >250 sec and or VWF:Act/VWF:Ag<0.7)
* Patient with a known thrombophilia
* Patient with a known severe bleeding disorder
* Patient refusal or environment
* Minor patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinically significant bleeding within 3 months after implantation | 3 months
  A clinically significant bleeding event is defined as internal or external bleeding leading to death or prolonged hospitalization or requiring re-hospitalization, surgery or transfusion of at least 3 units of packed red blood cells or hemoglobin drop> 3g/dL and/or refractory to conventional approach

CONTACTS AND LOCATIONS:
Overall Officials: Susen Sophie, MD, PhD, Study Chair — University Hospital, Lille
Locations (1):
- CHRU,, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincentelli A, Susen S, Le Tourneau T, Six I, Fabre O, Juthier F, Bauters A, Decoene C, Goudemand J, Prat A, Jude B. Acquired von Willebrand syndrome in aortic stenosis. N Engl J Med. 2003 Jul 24;349(4):343-9. doi: 10.1056/NEJMoa022831. PMID 12878741
- [Background] Van Belle E, Rauch A, Vincentelli A, Jeanpierre E, Legendre P, Juthier F, Hurt C, Banfi C, Rousse N, Godier A, Caron C, Elkalioubie A, Corseaux D, Dupont A, Zawadzki C, Delhaye C, Mouquet F, Schurtz G, Deplanque D, Chinetti G, Staels B, Goudemand J, Jude B, Lenting PJ, Susen S. Von Willebrand factor as a biological sensor of blood flow to monitor percutaneous aortic valve interventions. Circ Res. 2015 Mar 27;116(7):1193-201. doi: 10.1161/CIRCRESAHA.116.305046. Epub 2015 Feb 10. PMID 25670067